CLINICAL TRIAL: NCT02578147
Title: JUEGA: A Fun Study for Hispanic/Latino Adolescent Girls
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not available to continue enrollment beyond study completion date.
Sponsor: University of Miami (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Anne E. Norris, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20140697; R01NR014851 (NIH)
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Adolescent Behavior
Keywords: risky sexual behavior; early intervention; adolescent pregnancy
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mighty Girls (Experimental): Girls in this group complete 3 different activities after school: 6 classroom sessions, 4 DRAMA-RAMA game play sessions, and 4 short game experience surveys. Classroom sessions are 1 hour long, 3 days a week for 2 weeks. Topics include: goal setting, choices and their effects; defining what makes a behavior risky; learning how to not get talked into doing risky things by friends (e.g., going to a party at a house where parents are not home); and learning to be critical of TV shows and other media that make it seem like lots of teens are having sex. These sessions teach girls skills and strategies that help them score game points in DRAMA-RAMA. These are important skills and strategies that they can use in everyday life to make wise choices. Classroom sessions are designed to be fun.
  Interventions: Behavioral: Mighty Girls
- Game Girls (Active Comparator): Girls in this group take part in activities that can be done from home or anywhere they have Wi-Fi access: 4 Science Valley game play sessions and 4 short game experience surveys. Science Valley is a web based game in which girls explore a virtual world and experiment with objects in this world using a computer, tablet or cell phone. Girls will play this game for about 20-30 minutes. There are no classroom sessions required to be able to play Science Valley. Science Valley is designed to be fun and to give girls a chance to build skills important to doing well in school: her problem solving and critical thinking skills. Girls will be given a link to use to access Science Valley on the internet. At the end of the game, they do a short game experience survey that asks questions about how easy, how hard, how fun etc. it was to play Science Valley. This survey will appear on the screen at the end of the Science Valley game play session.
  Interventions: Behavioral: Game Girls

INTERVENTIONS:
Behavioral: Mighty Girls
  Arms: Mighty Girls
Behavioral: Game Girls
  Arms: Game Girls

SUMMARY:
The purpose of this study is to have girls play new computer games designed for middle school children and not yet available to the public. The investigator wants to know what girls think about these games. The investigator also wants to learn about the health behavior of 7th grade girls of Hispanic/Brazilian/Latino origin, and the investigators want to test the Mighty Girls program in Miami. Half of the girls in JUEGA will be given the Mighty Girls program and the investigators want to know if this program reduces behavior that puts girls at risk for having sex, drinking, and using drugs. The program tries to reduce this risk by helping girls learn skills to make wise choices, even when their friends have other ideas or want them to make more risky choices This goal is important because US statistics indicate that Hispanic teens are at risk for teen pregnancy and Miami has one of the highest HIV and AIDS rates in the United States. The investigator wants to find out whether the Mighty Girls program is as effective in Miami-Dade County Public Schools as it was when tested in one of Orlando's Orange County Public Schools.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* enrolled in 7th grade at a participating school

Exclusion Criteria:

* developmental delay

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 552 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in sexual intentions from baseline (pre-intervention) | baseline, 3 months, 12 months, 24 months
  Sexual intentions are defined as the change in a score from 1 (definitely not) to 4 (definitely yes) to engage in sexual intercourse in the near future on an electronic survey.
Change in risky sexual behavior from baseline (pre-intervention) | baseline, 3 months, 12 months, 24 months
  Risky sexual behavior is defined as the change in the percentage of participants reporting yes for engaging in heavy petting and percentage reporting yes for engaging in vaginal intercourse on an electronic survey.

SECONDARY OUTCOMES:
Change in sexual intentions from baseline (pre-intervention) as affected by the change in peer resistance self-efficacy | baseline, 3 months, 12 months, 24 months
  Peer resistance self-efficacy is defined as the change in a score from 1 (disagree strongly) to 4 (agree strongly) to resist peer pressure to engage in sexual behavior and/or put oneself at risk to be exposed to other teens engaging in risky sexual behavior on an electronic survey.
Change in sexual intentions from baseline (pre-intervention) as affected by implementation quality | baseline, 3 months, 12 months, 24 months
  Implementation quality is defined as the amount of participant engagement, intervener engagement, quality of intervener delivery, and content adherence (fidelity) on a score of 0 to 100.
Change in risky sexual behavior from baseline (pre-intervention) as affected by the change in peer resistance self-efficacy | baseline, 3 months, 12 months, 24 months
  Peer resistance self-efficacy is defined as the change in a score from 1 (disagree strongly) to 4 (agree strongly) to resist peer pressure to engage in sexual behavior and/or put oneself at risk to be exposed to other teens engaging in risky sexual behavior on electronic survey.
Change in risky sexual behavior from baseline (pre-intervention) as affected by implementation quality | baseline, 3 months, 12 months, 24 months
  Implementation quality is defined as the amount of participant engagement, intervener engagement, quality of intervener delivery, and content adherence (fidelity) on a score of 0 to 100.
Costs of implementation of the intervention | 4 months
  Costs of implementation are defined as participant transportation home from school intervention site; participant snacks; intervener salary (training, delivery, commuting time); intervention supplies, materials, and equipment; support from school personnel at the study site.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Norris, PhD, Principal Investigator — University of Miami
Locations (1):
- School of Nursing and Health Studies, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No